CLINICAL TRIAL: NCT00666809
Title: Evaluation of Vardenafil for the Treatment of Subjective Tinnitus: A Controlled Pilot Study
Brief Title: Vardenafil in Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12049; 2006-000463-29 (EudraCT Number)
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Tinnitus
Keywords: Vardenafil,; Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Vardenafil 10 mg BID p.o. for 12 weeks + 4 weeks follow-up
  Arms: Arm 1
Drug: Placebo — Placebo BID p.o. for 12 weeks + 4 weeks follow-up
  Arms: Arm 2

SUMMARY:
There is incidental evidence (casuistic findings) that the treatment with vardenafil of male patients suffering from erectile dysfunction and comorbid tinnitus experienced an improvement of their tinnitus.

Randomized, parallel-group, double-blind, placebo-controlled trial over 16 weeks (12 weeks of treatment + 4 weeks follow-up) with 10 mg vardenafil BID p.o. in men and women with chronic tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Chronic subjective cochlear tinnitus
* No treatment of tinnitus within 4 weeks prior to study entry
* Duration of tinnitus > 3 months

Exclusion Criteria:

* Acute tinnitus
* Intermittent tinnitus
* History of M. Menieré
* History of conductive deafness
* History of psychogenic deafness
* History of tumors of the middle ear, inner ear or cerebella-pontine angle (malignant and non malignant)
* Patients diagnosed of multiple sclerosis
* History of myocardial infarction, stroke, or life-threatening arrhythmia within the prior 6 months
* Nitrates or nitric oxide donors
* Any other concurrent treatment of tinnitus during study
* pregnant and breast-feeding women
* women with child-bearing potential not using adequate birth control method (Note: as adequate method of birth control oral contraception, spiral or sexual abstinence is recommended)
* Other exclusion criteria apply according to the Summary of Product Characteristics

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2006-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Total score of the Tinnitus | 4 times in 16 weeks

SECONDARY OUTCOMES:
Audiometric measurements (mode, frequency and loudness of tinnitus, pure tone audiogram, speech audiogram) | 16 weeks
Quality of life (SF 36 Questionnaire) | 16 weeks
Serum human chorionic Gonadotropin (hcG), pregnancy test | once at screening
Safety and tolerability | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, Berlin / 285, Germany

REFERENCES:
- See also: click here and search for Bayer product information provided by the EMA — http://www.clinicaltrialsregister.eu